CLINICAL TRIAL: NCT00811733
Title: A Phase II Trial of Ofatumumab in Subjects With Waldenstrom's Macroglobulinemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110921
Record Dates: First submitted 2008-12-18; First posted 2008-12-19 (Estimated); Results first posted 2012-04-30 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2015-03

CONDITIONS: Waldenstrom Macroglobulinaemia
Keywords: Waldenstrom's Macroglobulinemia; Ofatumumab
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — ofatumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ofatumumab (Experimental): Ofatumumab is a fully human antibody, targeting a unique epitope on the CD20 molecule expressed on human B cells.
  Interventions: Biological: Ofatumumab

INTERVENTIONS:
Biological: Ofatumumab — Ofatumumab is a fully human antibody, targeting a unique epitope on the CD20 molecule expressed on human B cells.

SUMMARY:
Given the tolerability and efficacy of ofatumumab in follicular lymphoma and Chronic Lymphocytic Leukemia, and the need to improve therapy for patients with WM utilizing a non-myelosuppressive agent this phase II trial of ofatumumab is being initiated in patients with Waldenstrom's Macroglobulinemia (WM).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed and active Waldenstrom's Macroglobulinemia requiring treatment.
* Ambulatory and capable of all selfcare. Up and about more than 50% of waking hours.
* Adequate organ function.
* Detectable CD20 positive of the tumor cells.
* Measurable disease as defined by a monoclonal IgM paraprotein level greater than 1000 mg/dL.

Exclusion Criteria:

* Treatment of WM within the past 28 days.
* Treatment with rituximab or alemtuzamab within the past 3 months.
* Certain heart problems, chronic or current active infection not controlled with oral antibiotics, other current cancer or within last 5 years.
* Current participation in another interventional clinical study.
* Lactating or pregnant women or female patients of child-bearing potential (or male patients with such partners) not willing to use adequate contraception.
* Active cerebrovascular disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2009-03-01; Primary Completion 2011-06-01 (Actual); Study Completion 2014-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- United States (7):
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Stanford, California
  - GSK Investigational Site, Rochester, Minnesota
  - GSK Investigational Site, Buffalo, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, San Antonio, Texas

REFERENCES:
- [Derived] Furman RR, Eradat HA, DiRienzo CG, Hofmeister CC, Hayman SR, Leonard JP, Coleman M, Advani R, Chanan-Khan A, Switzky J, Liao QM, Shah D, Jewell RC, Lisby S, Lin TS. Once-weekly ofatumumab in untreated or relapsed Waldenstrom's macroglobulinaemia: an open-label, single-arm, phase 2 study. Lancet Haematol. 2017 Jan;4(1):e24-e34. doi: 10.1016/S2352-3026(16)30166-1. Epub 2016 Dec 1. PMID 27914971

RESULTS

PARTICIPANT FLOW:
Groups:
- 300 mg Ofatumumab, Wk. 1; 1000/2000 mg Ofatumumab, Wk. 2-4/2-5: Participants received ofatumumab intravenously (IV) in Cycle 1 (defined as a treatment period of up to 4 weeks [Weeks (Wk.) 1 through 4]) (300 milligrams [mg] at Week 1 and 1000 mg at Weeks 2 through 4) and were followed up for 11 weeks (Weeks 5-16). After Week 16, during the Redosing Cycle (RC), participants who had Minor Response or stable disease after Cycle 1 and had not received another Waldenstrom's Macroglobulinemia (WM) therapy received 300 mg IV ofatumumab at Week 1 and 2000 mg IV ofatumumab at Weeks 2 through 5. Participants who achieved a response in either Cycle 1 or the RC and subsequently progressed before 36 months entered Cycle 2 of treatment and received IV ofatumumab 300 mg at Week 1 and IV ofatumumab 2000 mg during Weeks 2 through 5.
- 300 mg Ofatumumab, Wk. 1; 2000 mg Ofatumumab, Wk. 2-5: Participants received ofatumumab IV at 300 mg at Week 1 and 2000 mg at Weeks 2 through 5 in Cycle 1 (defined as a treatment period of up to 5 weeks [Weeks 1 through 5]) and were followed up for 10 weeks (Weeks 6-16). After Week 16, during the RC, participants who had Minor Response or stable disease after Cycle 1 and had not received another WM therapy received 300 mg IV ofatumumab at Week 1 and 2000 mg IV ofatumumab at Weeks 2 through 5. Participants who achieved a response and subsequently progressed before 36 months entered Cycle 2 of treatment and received 300 mg at Week 1 and 2000 mg during Weeks 2 through 5.
Period: Overall Study
Arm/Group | 300 mg Ofatumumab, Wk. 1; 1000/2000 mg Ofatumumab, Wk. 2-4/2-5 | 300 mg Ofatumumab, Wk. 1; 2000 mg Ofatumumab, Wk. 2-5
Started | 15 | 22
Completed | 4 | 12
Not Completed | 11 | 10
Not completed — Investigator Discretion | 10 | 8
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 300 mg Ofatumumab, Wk. 1; 1000/2000 mg Ofatumumab, Wk. 2-4/2-5 | 300 mg Ofatumumab, Wk. 1; 2000 mg Ofatumumab, Wk. 2-5 | Total
Number analyzed (Participants) | 15 | 22 | 37
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.3 (10.78) | 64.0 (9.36) | 63.3 (9.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 15
  Male | 9 | 13 | 22
Race/Ethnicity, Customized [Number; unit: participants]
  African American/African Heritage | 0 | 1 | 1
  Asian - East Asian Heritage | 0 | 1 | 1
  White - White/Caucasian/European | 14 | 19 | 33
  Unknown | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Overall Response (OR) for Cycle 1 (Including the Redosing Cycle), as Assessed by the Investigator
Description: OR (based on the Consensus Panel recommendations from the 2nd and 3rd International Workshop on WM) included Complete Response (CR), Partial Response (PR), or a Minor Response (MR). CR: Complete disappearance of serum monoclonal (SM) Immunoglobulin (Ig) E (IgE), measured centrally; resolution of adenopathy/organomegaly upon physical exam and computerized tomography (CT) scan; lymph nodes =<1.5 centimeters; absence of malignant cell by bone marrow histologic examination. PR: a >=50% reduction from baseline in the SM IgM concentration. MR: >=25%, but a <50% reduction of SM IgM from baseline.
Time Frame: Baseline and up to 27 months from the first dose of Cycle 1 (Study Day 1), and before Cycle 2 treatment
Population: Intent-to-Treat (ITT) Population: all participants who were considered eligible for treatment and who had been exposed to study drug irrespective of the planned course of treatment.
Measure: Number; unit: participants
Arm/Group | 300 mg Ofatumumab, Wk. 1; 1000/2000 mg Ofatumumab, Wk. 2-4/2-5 | 300 mg Ofatumumab, Wk. 1; 2000 mg Ofatumumab, Wk. 2-5
Number analyzed (Participants) | 15 | 22
participants | 7 | 15
Statistical Analysis 1: Comparison: 300 mg Ofatumumab, Wk. 1; 1000/2000 mg Ofatumumab, Wk. 2-4/2-5; Test type: Superiority or Other; percentage of participants = 47, 95% CI 2-sided [21.3 to 73.4] — The estimated value represents the percentage of participants with OR
Statistical Analysis 2: Comparison: 300 mg Ofatumumab, Wk. 1; 2000 mg Ofatumumab, Wk. 2-5; Test type: Superiority or Other; percentage of participants = 68, 95% CI 2-sided [45.1 to 86.1] — The estimated value represents the percentage of participants with OR

2. Primary Outcome: Number of Participants With OR for Cycle 1 (Excluding the Redosing Cycle), as Assessed by the Investigator
Description: as for outcome 1
Time Frame: Baseline and up to Study Week 16
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | 300 mg Ofatumumab, Wk. 1; 1000/2000 mg Ofatumumab, Wk. 2-4/2-5 | 300 mg Ofatumumab, Wk. 1; 2000 mg Ofatumumab, Wk. 2-5
Number analyzed (Participants) | 15 | 22
participants | 5 | 14
Statistical Analysis 1: Comparison: 300 mg Ofatumumab, Wk. 1; 1000/2000 mg Ofatumumab, Wk. 2-4/2-5; Test type: Superiority or Other; percentage of participants = 33, 95% CI 2-sided [11.8 to 61.6] — The estimated value represents the percentage of participants with OR
Statistical Analysis 2: Comparison: 300 mg Ofatumumab, Wk. 1; 2000 mg Ofatumumab, Wk. 2-5; Test type: Superiority or Other; percentage of participants = 64, 95% CI 2-sided [40.7 to 82.8] — The estimated value represents the percentage of participants with OR

3. Secondary Outcome: Number of Participants With CR, PR, and MR for Cycle 1 (Including the Redosing Cycle), as Assessed by the Investigator
Description: Response criteria were based on the Consensus Panel recommendations from the 2nd and 3rd International Workshop on WM. CR: Complete disappearance of serum monoclonal (SM) Immunoglobulin (Ig) E (IgE), measured centrally; resolution of adenopathy/organomegaly upon physical exam and computerized tomography (CT) scan; lymph nodes =<1.5 centimeters; absence of malignant cell by bone marrow histologic examination. PR: a >=50% reduction from baseline in the SM IgM concentration. MR: >=25%, but a <50% reduction of SM IgM from baseline.
Time Frame: Baseline and up to 27 months from the first dose of Cycle 1 (Study Day 1), and before Cycle 2 treatment
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | 300 mg Ofatumumab, Wk. 1; 1000/2000 mg Ofatumumab, Wk. 2-4/2-5 | 300 mg Ofatumumab, Wk. 1; 2000 mg Ofatumumab, Wk. 2-5
Number analyzed (Participants) | 15 | 22
participants
  CR | 0 | 0
  PR | 4 | 11
  MR | 3 | 4

4. Secondary Outcome: Number of Participants With CR, PR, and MR for Cycle 1 (Excluding the Redosing Cycle), as Assessed by the Investigator
Description: as for outcome 3
Time Frame: Baseline and up to Study Week 16
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | 300 mg Ofatumumab, Wk. 1; 1000/2000 mg Ofatumumab, Wk. 2-4/2-5 | 300 mg Ofatumumab, Wk. 1; 2000 mg Ofatumumab, Wk. 2-5
Number analyzed (Participants) | 15 | 22
participants
  CR | 0 | 0
  PR | 3 | 9
  MR | 2 | 5

5. Secondary Outcome: Number of Participants With IgM Flare for Cycle 1 Response (Including the Redosing Cycle)
Description: IgM is a basic antibody that is produced by B cells. It is the first antibody to appear in response to initial exposure to antigen. IgM flare is defined as an IgM level that increases by >25% from baseline (BL) and is associated with a response to treatment. Avoidance of IgM flare indicates the lack of an increase in IgM of >25% from BL.
Time Frame: Baseline and up to 27 months from the first dose of Cycle 1 (Study Day 1), and before Cycle 2 treatment
Population: ITT Population. Only those participants who received Cycle 1 treatment (including the Redosing Cycle) were assessed.
Measure: Number; unit: participants
Arm/Group | 300 mg Ofatumumab, Wk. 1; 1000/2000 mg Ofatumumab, Wk. 2-4/2-5 | 300 mg Ofatumumab, Wk. 1; 2000 mg Ofatumumab, Wk. 2-5
Number analyzed (Participants) | 15 | 22
participants
  >25% increase from BL, any response, n=15, 22 | 7 | 9
  =<25% increase from BL, any response, n=15, 22 | 8 | 13
  >25% increase from BL, PR/MR response , n=7, 15 | 1 | 2
  =<25% increase from BL, PR/MR response , n=7, 15 | 6 | 13

6. Secondary Outcome: Duration of Response for All Responders (CR, PR, MR), as Assessed by the Investigator
Description: Duration of response is defined as the time from the initial response to relapse/disease progression (DP) or death. DP for CR is defined as the reappearance of the IgM protein, new signs/symptoms attributable to WM, evidence of active disease or recurrence of bone marrow involvement by lymphoplasmacytic cells, or the appearance of any new lymph node >=1.5 centimeters on any axis. Progression for PR/MR is either a >=25% increase in IgM from the lowest attained response value or progression of lymphadenopathy, organomegaly, cytopenias, or other clinically significant signs/symptoms caused by WM.
Time Frame: From baseline up to approximately 5 years
Population: ITT Population. Only those participants classified as responders were included in the analysis. Participants who had disease progression or death were counted as events, and other participants were censored at the date of the last adequate assessment in the study.
Measure: Median (Inter-Quartile Range); unit: days
Units Other Than Participants: events
Arm/Group | 300 mg Ofatumumab, Wk. 1; 1000/2000 mg Ofatumumab, Wk. 2-4/2-5 | 300 mg Ofatumumab, Wk. 1; 2000 mg Ofatumumab, Wk. 2-5
Number analyzed (Participants) | 7 | 15
Number analyzed (events) | 5 | 9
days | 449.0 [275.0 to NA] — There were too few events (disease progression or death) to estimate the third quartile. | 455.0 [337.0 to 1016.0]

7. Secondary Outcome: Progression-free Survival
Description: Time to disease progression is defined as the time from baseline to disease progression or death.
Time Frame: From baseline up to approximately 5 years
Population: ITT Population. Participants who experienced disease progression or death were counted as events, and other participants were censored at the time of the last adequate assessment in the study.
Measure: Median (Inter-Quartile Range); unit: days
Units Other Than Participants: events
Arm/Group | 300 mg Ofatumumab, Wk. 1; 1000/2000 mg Ofatumumab, Wk. 2-4/2-5 | 300 mg Ofatumumab, Wk. 1; 2000 mg Ofatumumab, Wk. 2-5
Number analyzed (Participants) | 15 | 22
Number analyzed (events) | 8 | 13
days | 558.0 [353.0 to 666.0] | 536.0 [414.0 to 1093.0]

8. Secondary Outcome: Time to Response for Responders
Description: Time to response is defined as the time from baseline to the first response date.
Time Frame: From baseline up to approximately 5 years
Population: ITT Population. Only participants classified as responders (CR, PR, and MR) were assessed.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | 300 mg Ofatumumab, Wk. 1; 1000/2000 mg Ofatumumab, Wk. 2-4/2-5 | 300 mg Ofatumumab, Wk. 1; 2000 mg Ofatumumab, Wk. 2-5
Number analyzed (Participants) | 7 | 15
days | 78 [72 to 269] | 81 [78 to 104]

9. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from baseline until death due to any cause.
Time Frame: From baseline up to approximately 5 years
Population: ITT Population. Only those participants who died during the study and during the follow-up period were assessed.
Arm/Group | 300 mg Ofatumumab, Wk. 1; 1000/2000 mg Ofatumumab, Wk. 2-4/2-5 | 300 mg Ofatumumab, Wk. 1; 2000 mg Ofatumumab, Wk. 2-5
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Clearance of Ofatumumab
Description: Clearance (CL) is defined as the volume of plasma that is cleared of drug per unit of time. Blood samples for the quantification of ofatumumab were collected during each cycle and for up to 6 months after the end of each cycle.
Time Frame: From the first dose (Cycle 1 Day 1) up to 6 months after the end of the last cycle of treatment; blood collected on each dosing day, weekly up to Week 8, and every 4 weeks up to Week 24/Month 7
Population: Pharmacokinetic (PK) Population: all participants from whom a PK sample was obtained and analyzed. Data were provided for the number of participants for whom the parameter could be determined.
Measure: Geometric Mean (95% Confidence Interval); unit: milliliters/hour (ml/hr)
Arm/Group | 300 mg Ofatumumab, Wk. 1; 1000/2000 mg Ofatumumab, Wk. 2-4/2-5 | 300 mg Ofatumumab, Wk. 1; 2000 mg Ofatumumab, Wk. 2-5
Number analyzed (Participants) | 15 | 21
milliliters/hour (ml/hr) | 27.9 [16.0 to 48.6] | 13.5 [8.7 to 20.8]

11. Secondary Outcome: Volume of Distribution at Steady State of Ofatumumab
Description: Volume of distribution at steady state (Vss) is defined as the apparent volume of distribution of the drug in the body at steady state. Blood samples for the quantification of ofatumumab were collected during each cycle and for up to 6 months after the end of each cycle.
Time Frame: as for outcome 10
Population: PK Population. Data were provided for the number of participants for whom the parameter could be determined.
Measure: Geometric Mean (95% Confidence Interval); unit: Liters (L)
Arm/Group | 300 mg Ofatumumab, Wk. 1; 1000/2000 mg Ofatumumab, Wk. 2-4/2-5 | 300 mg Ofatumumab, Wk. 1; 2000 mg Ofatumumab, Wk. 2-5
Number analyzed (Participants) | 15 | 21
Liters (L) | 10.0 [8.9 to 11.2] | 10.7 [9.6 to 12.0]

12. Secondary Outcome: Half-life of Ofatumumab
Description: Half-life (t½) is defined as the time required for the concentration of the drug in plasma to decrease to one-half of its current value. Blood samples for the quantification of ofatumumab were collected during each cycle and for up to 6 months after the end of each cycle.
Time Frame: as for outcome 10
Population: PK Population. Data were provided for the number of participants for whom the parameter could be determined.
Measure: Geometric Mean (95% Confidence Interval); unit: Days (d)
Arm/Group | 300 mg Ofatumumab, Wk. 1; 1000/2000 mg Ofatumumab, Wk. 2-4/2-5 | 300 mg Ofatumumab, Wk. 1; 2000 mg Ofatumumab, Wk. 2-5
Number analyzed (Participants) | 15 | 21
Days (d) | 10.9 [6.8 to 17.5] | 23.9 [16.2 to 35.2]

13. Secondary Outcome: Cmax and Ctrough of Ofatumumab
Description: Cmax is defined as the maximum observed drug concentration after administration, and Ctrough is defined as the drug concentration observed prior to the start of the next dose. Blood samples for the quantification of ofatumumab were collected during each cycle and for up to 6 months after the end of each cycle.
Time Frame: as for outcome 10
Population: PK Population. Data were provided for the number of participants attending each visit for whom the parameter could be determined.
Measure: Geometric Mean (95% Confidence Interval); unit: micrograms/milliliter (µg/ml)
Arm/Group | 300 mg Ofatumumab, Wk. 1; 1000/2000 mg Ofatumumab, Wk. 2-4/2-5 | 300 mg Ofatumumab, Wk. 1; 2000 mg Ofatumumab, Wk. 2-5
Number analyzed (Participants) | 15 | 21
micrograms/milliliter (µg/ml)
  Cmax, Course 1 Dose 1, n=14,19 | 68.3 [48.0 to 97.1] | 72.1 [57.4 to 90.6]
  Cmax, Course 1 Dose 3, n=0,19 | NA [NA to NA] — No participants were analyzed at the indicated time point; therefore, the mean and the CI could not be calculated. | 465 [386 to 561]
  Cmax, Course 1 Dose 4, n=13,0 | 259 [195 to 344] | NA [NA to NA] — No participants were analyzed at the indicated time point; therefore, the mean and the CI could not be calculated.
  Cmax, Course 1 Dose 5, n=0,18 | NA [NA to NA] — No participants were analyzed at the indicated time point; therefore, the mean and the CI could not be calculated. | 640 [523 to 783]
  Ctrough, Course 1 Dose 2, n=7,12 | 3.0 [0.3 to 27.4] | 8.0 [2.0 to 32.2]
  Ctrough, Course 1 Dose 3, n=11,19 | 13.9 [2.1 to 91.3] | 121 [67.3 to 217]
  Ctrough, Course 1 Dose 4, n=13,21 | 23.4 [4.3 to 128] | 181 [95.3 to 344]
  Ctrough, Course 1 Dose 5, n=0,18 | NA [NA to NA] — No participants were analyzed at the indicated time point; therefore, the mean and the CI could not be calculated. | 249 [127 to 489]
  Cmax, Course 2 Dose 1, n=9,11 | 53.2 [33.1 to 85.6] | 64.8 [42.8 to 98.2]
  Cmax, Course 2 Dose 3, n=8,12 | 554 [420 to 730] | 577 [436 to 762]
  Cmax, Course 2 Dose 5, n=10,12 | 528 [339 to 825] | 803 [616 to 1046]
  Ctrough, Course 2 Dose 2, n=7,10 | 8.1 [1.2 to 52.7] | 20.4 [4.7 to 89.2]
  Ctrough, Course 2 Dose 3, n=8,12 | 144 [64.6 to 319] | 169 [102 to 280]
  Ctrough, Course 2 Dose 4, n=11,12 | 225 [110 to 458] | 310 [200 to 482]
  Ctrough, Course 2 Dose 5, n=11,12 | 279 [155 to 503] | 384 [273 to 542]

14. Secondary Outcome: AUC(0-tau) and AUC(0-inf) of Ofatumumab
Description: AUC(0-tau) is the area under the drug concentration-time curve over the dosing interval (one week). AUC(0-inf) is the area under the drug concentration-time curve from time zero extrapolated to infinite time. Blood samples for the quantification of ofatumumab were collected during each cycle and for up to 6 months after the end of each cycle.
Time Frame: as for outcome 10
Population: PK Population. Data were provided for the number of participants attending each visit for whom the parameter could be calculated..
Measure: Geometric Mean (95% Confidence Interval); unit: micrograms X hours/milliliters (µg.h/mL)
Arm/Group | 300 mg Ofatumumab, Wk. 1; 1000/2000 mg Ofatumumab, Wk. 2-4/2-5 | 300 mg Ofatumumab, Wk. 1; 2000 mg Ofatumumab, Wk. 2-5
Number analyzed (Participants) | 15 | 21
micrograms X hours/milliliters (µg.h/mL)
  AUC(0-tau), Course 1 Dose 4, n=13,0 | 21419 [11637 to 39424] | NA [NA to NA] — No participants were analyzed at the indicated time point; therefore, the mean and the CI could not be calculated.
  AUC(0-tau), Course 1 Dose 5, n=0,18 | NA [NA to NA] — No participants were analyzed at the indicated time point; therefore, the mean and the CI could not be calculated. | 75526 [56462 to 101028]
  AUC(0-inf), Course 1 Dose 4, n=9,0 | 120886 [53956 to 270842] | NA [NA to NA] — No participants were analyzed at the indicated time point; therefore, the mean and the CI could not be calculated.
  AUC(0-inf), Course 1 Dose 5, n=0,18 | NA [NA to NA] — No participants were analyzed at the indicated time point; therefore, the mean and the CI could not be calculated. | 392012 [220019 to 698454]
  AUC(0-tau), Course 2 Dose 5, n=10,12 | 61259 [36684 to 102296] | 106275 [82044 to 137663]
  AUC(0-inf), Course 2 Dose 5, n=8,12 | 221675 [70622 to 695814] | 507794 [286020 to 901528]

15. Secondary Outcome: Number of Participants With at Least One Confirmed Positive Post-ofatumumab HAHA Result
Description: All human-antihuman antibody (HAHA) samples were first tested in a screening assay to identify potential HAHA positives. Next, samples that tested positive in the screening assay were further tested in the confirmation assay to determine the specificity of the signal to ofatumumab. Confirmed positive samples were reported as positive.
Time Frame: From baseline up to approximately 5 years
Population: Safety Population. Only those participants with post-ofatumumab HAHA results were analyzed.
Measure: Number; unit: participants
Arm/Group | 300 mg Ofatumumab, Wk. 1; 1000/2000 mg Ofatumumab, Wk. 2-4/2-5 | 300 mg Ofatumumab, Wk. 1; 2000 mg Ofatumumab, Wk. 2-5
Number analyzed (Participants) | 11 | 20
participants | 1 | 4

16. Secondary Outcome: Change From Baseline in Blood Counts (CD4+, CD19+, CD50) at Month 3 After Treatment
Description: CD4+ and CD19+ are two key flow cytometry parameters, and total hemolytic complement (CD50) is a complement parameter. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and Month 3
Population: ITT Population: only participants with blood count data at both Baseline and Month 3 were included in the analysis.
Measure: Median (Full Range); unit: cells per microliter (µL)
Arm/Group | 300 mg Ofatumumab, Wk. 1; 1000/2000 mg Ofatumumab, Wk. 2-4/2-5 | 300 mg Ofatumumab, Wk. 1; 2000 mg Ofatumumab, Wk. 2-5
Number analyzed (Participants) | 15 | 22
cells per microliter (µL)
  CD4+ | -35.5 [-277 to 194] | 98 [-50 to 503]
  CD19+ | -26 [-734 to 0] | -24.5 [-61 to -9]
  CD50 | 9 [-122 to 104] | -43 [-287 to 50]

17. Secondary Outcome: Number of Participants With the Indicated SAEs Related to Study Drug
Description: An SAE is any event occurring at any dose that results in any of the following: death, a life-threatening adverse drug experience (ADE; at immediate risk of death from the experience as it occurred), inpatient hospitalization/prolongation of existing hospitalization, a persistent/significant disability/incapacity, or a congenital anomaly/birth defect. Medical events that may not result in death, be life threatening, or require hospitalization may be considered to be a serious ADEs when based upon appropriate medical judgment. Relatedness was based on the Investigator's medical judgement.
Time Frame: From baseline up to approximately 5 years
Population: Safety Population. Only those participants who experienced an SAE categorized as being related to study drug were assessed.
Measure: Number; unit: participants
Arm/Group | 300 mg Ofatumumab, Wk. 1; 1000/2000 mg Ofatumumab, Wk. 2-4/2-5 | 300 mg Ofatumumab, Wk. 1; 2000 mg Ofatumumab, Wk. 2-5
Number analyzed (Participants) | 2 | 2
participants
  Haemolysis | 0 | 1
  Chest pain | 0 | 1
  Cryoglobulinaemia | 1 | 0
  Fluid overload | 0 | 1
  Renal failure acute | 1 | 0
  Pulmonary oedema | 0 | 1

18. Secondary Outcome: Number of Participants With the Indicated SAEs and Non-serious AEs Related to Study Drug
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. The Investigator assessed whether the AE was possibly or probably related to study drug.
Time Frame: From baseline up to approximately 5 years
Population: Safety Population. Only those participants who experienced a study drug-related AE were assessed.
Measure: Number; unit: participants
Arm/Group | 300 mg Ofatumumab, Wk. 1; 1000/2000 mg Ofatumumab, Wk. 2-4/2-5 | 300 mg Ofatumumab, Wk. 1; 2000 mg Ofatumumab, Wk. 2-5
Number analyzed (Participants) | 13 | 22
participants
  Pruritus | 4 | 8
  Urticaria | 4 | 9
  Rash | 4 | 3
  Pruritus generalised | 2 | 1
  Hyperhidrosis | 1 | 1
  Erythema | 1 | 0
  Palmar erythema | 0 | 1
  Rash macular | 1 | 0
  Swelling face | 0 | 1
  Throat irritation | 7 | 3
  Nasal congestion | 1 | 2
  Oropharyngeal pain | 0 | 3
  Dyspnoea | 0 | 1
  Epistaxis | 0 | 1
  Painful respiration | 0 | 1
  Pulmonary oedema | 0 | 1
  Rhinitis allergic | 0 | 1
  Rhinorrhoea | 1 | 0
  Sneezing | 0 | 1
  Pyrexia | 2 | 5
  Chills | 1 | 5
  Chest pain | 1 | 1
  Chest discomfort | 2 | 0
  Fatigue | 1 | 2
  Non-cardiac chest pain | 2 | 0
  Asthenia | 0 | 1
  Ill-defined disorder | 1 | 0
  Local swelling | 0 | 1
  Malaise | 0 | 1
  Pain | 1 | 0
  Abdominal pain | 2 | 1
  Diarrhoea | 0 | 3
  Nausea | 0 | 2
  Paraesthesia oral | 0 | 2
  Abdominal discomfort | 1 | 0
  Dyspepsia | 1 | 0
  Hypoaesthesia oral | 0 | 1
  Lip swelling | 1 | 0
  Oral pain | 0 | 1
  Oral pruritus | 0 | 1
  Stomatitis | 0 | 1
  Flushing | 6 | 4
  Hypotension | 0 | 1
  Back pain | 1 | 1
  Limb discomfort | 0 | 1
  Muscle spasms | 1 | 0
  Musculoskeletal pain | 1 | 0
  Myalgia | 0 | 2
  Trismus | 1 | 0
  Anaemia | 0 | 2
  Haemolysis | 1 | 1
  Leukopenia | 0 | 1
  Lymph node pain | 1 | 0
  Neutropenia | 0 | 1
  Ear pruritus | 3 | 2
  Eye pruritus | 3 | 0
  Ocular hyperaemia | 1 | 1
  Abnormal sensation in eye | 0 | 1
  Eye swelling | 0 | 1
  Decreased appetite | 2 | 1
  Fluid overload | 0 | 1
  Hypophagia | 0 | 1
  Increased appetite | 0 | 1
  Headache | 1 | 1
  Paraesthesia | 0 | 2
  Sinus headache | 1 | 0
  Infusion related reaction | 2 | 3
  Blood creatinine increased | 1 | 0
  Body temperature increased | 0 | 1
  Protein total increased | 0 | 1
  Hypersensitivity | 0 | 1
  Serum sickness | 1 | 0
  Rhinitis | 1 | 0
  Urinary tract infection | 0 | 1
  Bradycardia | 1 | 0
  Insomnia | 0 | 1
  Renal failure acute | 1 | 0
  Thirst | 1 | 0
  Vomiting | 0 | 1
  Cryoglobulinaemia | 1 | 0
  Pallor | 1 | 0
  Arthralgia | 1 | 1
  Fluid retention | 1 | 0
  Hypoaesthesia | 0 | 1
  Psychomotor hyperactivity | 0 | 1
  Weight decreased | 1 | 0

19. Secondary Outcome: Number of Participants With the Indicated AEs Leading to Permanent Discontinuation of Study Drug and Withdrawal From Study
Description: Certain AEs led to permanent discontinuation of study drug and hence resulted in their withdrawal from the study.
Time Frame: From baseline up to approximately 5 years
Population: Safety Population. Only those participants who experienced an AE leading to their withdrawal from the study were assessed.
Measure: Number; unit: participants
Arm/Group | 300 mg Ofatumumab, Wk. 1; 1000/2000 mg Ofatumumab, Wk. 2-4/2-5 | 300 mg Ofatumumab, Wk. 1; 2000 mg Ofatumumab, Wk. 2-5
Number analyzed (Participants) | 2 | 1
participants
  Haemolysis | 1 | 1
  Febrile neutropenia | 1 | 0
  Myocardial ischaemia | 0 | 1
  Fluid overload | 0 | 1
  Renal failure acute | 1 | 0
  Pulmonary oedema | 0 | 1
  Haemolytic anaemia | 0 | 1

20. Secondary Outcome: Number of Participants With the Indicated >=Grade 3 AEs
Description: AEs were graded using the Common Toxicity Criteria for AEs from the Cancer Therapy Evaluation Program, Division of Cancer Therapy, National Cancer Institute. Grades: 0 = No AE or within normal limits; 1 = Mild AE; 2 = Moderate AE; 3 = Severe and undesirable AE; 4 = Life-threatening or disabling AE; 5 = Death related to AE.
Time Frame: From baseline up to approximately 5 years
Population: Safety Population. Only those participants who experienced a >=Grade 3 AE were assessed.
Measure: Number; unit: participants
Arm/Group | 300 mg Ofatumumab, Wk. 1; 1000/2000 mg Ofatumumab, Wk. 2-4/2-5 | 300 mg Ofatumumab, Wk. 1; 2000 mg Ofatumumab, Wk. 2-5
Number analyzed (Participants) | 8 | 8
participants
  Haemolysis | 1 | 1
  Anaemia | 1 | 0
  Febrile neutropenia | 1 | 0
  Haemolytic anaemia | 0 | 1
  Chest pain | 1 | 1
  Chest discomfort | 1 | 0
  Pyrexia | 0 | 1
  Blood creatinine increased | 1 | 0
  Haemoglobin decreased | 0 | 1
  Protein total increased | 0 | 1
  Dyspnoea exertional | 0 | 1
  Epistaxis | 1 | 0
  Pulmonary oedema | 0 | 1
  Cryoglobulinaemia | 1 | 0
  Serum sickness | 1 | 0
  Dizziness | 0 | 1
  Headache | 1 | 0
  Syncope | 0 | 1
  Myocardial ischaemia | 0 | 1
  Abdominal discomfort | 1 | 0
  Urinary tract infection | 0 | 1
  Fluid overload | 0 | 1
  Back pain | 0 | 1
  Renal failure acute | 1 | 0
  Rash | 1 | 0
  Neutropenia | 1 | 1
  Fatigue | 0 | 1
  Small intestinal obstruction | 0 | 1

21. Secondary Outcome: Number of Participants With the Indicated Infusion-related >=Grade 3 AE
Description: Infusion-related AEs are the AEs that resulted from administration of study drug through infusion. AEs were graded using the Common Toxicity Criteria for AEs from the Cancer Therapy Evaluation Program, Division of Cancer Therapy, National Cancer Institute. Grades: 0 = No AE or within normal limits; 1 = Mild AE; 2 = Moderate AE; 3 = Severe and undesirable AE; 4 = Life-threatening or disabling AE; 5 = Death related to AE.
Time Frame: From baseline up to approximately 5 years
Population: Safety Population. Only those participants who experienced >=Grade 3 infusion-related AEs were assessed.
Measure: Number; unit: participants
Arm/Group | 300 mg Ofatumumab, Wk. 1; 1000/2000 mg Ofatumumab, Wk. 2-4/2-5 | 300 mg Ofatumumab, Wk. 1; 2000 mg Ofatumumab, Wk. 2-5
Number analyzed (Participants) | 2 | 2
participants
  Chest pain | 1 | 1
  Chest discomfort | 1 | 0
  Back pain | 0 | 1
  Rash | 1 | 0

ADVERSE EVENTS:
Time Frame: Participants were followed from baseline up to approximately 5 years.
Arm/Group | 300 mg Ofatumumab, Wk. 1; 1000/2000 mg Ofatumumab, Wk. 2-4/2-5 | 300 mg Ofatumumab, Wk. 1; 2000 mg Ofatumumab, Wk. 2-5
Serious Adverse Events (participants affected / at risk) | 5/15 | 7/22
Other Adverse Events (participants affected / at risk) | 15/15 | 20/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 300 mg Ofatumumab, Wk. 1; 1000/2000 mg Ofatumumab, Wk. 2-4/2-5 (N=15) | 300 mg Ofatumumab, Wk. 1; 2000 mg Ofatumumab, Wk. 2-5 (N=22)
Catheter site haemorrhage (General disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 2
Haemolysis (Blood and lymphatic system disorders) | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 1 | 0
Cryoglobulinaemia (Immune system disorders) | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 300 mg Ofatumumab, Wk. 1; 1000/2000 mg Ofatumumab, Wk. 2-4/2-5 (N=15) | 300 mg Ofatumumab, Wk. 1; 2000 mg Ofatumumab, Wk. 2-5 (N=22)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 7 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 8
Urticaria (Skin and subcutaneous tissue disorders) | 4 | 9
Rash (Skin and subcutaneous tissue disorders) | 6 | 3
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 | 0
Nail bed bleeding (Skin and subcutaneous tissue disorders) | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0
Pyrexia (General disorders) | 3 | 5
Fatigue (General disorders) | 4 | 4
Chills (General disorders) | 1 | 5
Asthenia (General disorders) | 0 | 3
Chest pain (General disorders) | 1 | 2
Chest discomfort (General disorders) | 2 | 0
Non-cardiac chest pain (General disorders) | 2 | 0
Oedema (General disorders) | 0 | 2
Oedema peripheral (General disorders) | 2 | 0
Ill-defined disorder (General disorders) | 1 | 0
Medical device pain (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 2
Constipation (Gastrointestinal disorders) | 2 | 2
Diarrhea (Gastrointestinal disorders) | 2 | 3
Dyspepsia (Gastrointestinal disorders) | 2 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 2
Paraesthesia oral (Gastrointestinal disorders) | 0 | 2
Stomatitis (Gastrointestinal disorders) | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Lip swelling (Gastrointestinal disorders) | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Headache (Nervous system disorders) | 5 | 4
Paraesthesia (Nervous system disorders) | 1 | 3
Dizziness (Nervous system disorders) | 1 | 2
Hypoaesthesia (Nervous system disorders) | 1 | 2
Tremor (Nervous system disorders) | 1 | 1
Polyneuropathy (Nervous system disorders) | 1 | 0
Restless legs syndrome (Nervous system disorders) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 7 | 2
Sinusitis (Infections and infestations) | 2 | 3
Urinary tract infection (Infections and infestations) | 3 | 1
Nasopharyngitis (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 2 | 0
Bronchitis (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2
Iron deficiency (Metabolism and nutrition disorders) | 1 | 1
Haemochromatosis (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 4
Depression (Psychiatric disorders) | 1 | 0
Libido decreased (Psychiatric disorders) | 1 | 0
Flushing (Vascular disorders) | 6 | 4
Hot flush (Vascular disorders) | 1 | 0
Pallor (Vascular disorders) | 1 | 0
Raynaud's phenomenon (Vascular disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Trismus (Musculoskeletal and connective tissue disorders) | 1 | 0
Ear pruritus (Ear and labyrinth disorders) | 3 | 3
Deafness (Ear and labyrinth disorders) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Blood parathyroid hormone increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Eye pruritus (Eye disorders) | 3 | 0
Ocular hyperaemia (Eye disorders) | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 3
Palpitations (Cardiac disorders) | 1 | 1
Bradycardia (Cardiac disorders) | 1 | 0
Seasonal allergy (Immune system disorders) | 1 | 0
Serum sickness (Immune system disorders) | 1 | 0
Von Willebrand's disease (Congenital, familial and genetic disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Thirst (General disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Tongue ulceration (Gastrointestinal disorders) | 1 | 0
Candida infection (Infections and infestations) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 2
Sinus headache (Nervous system disorders) | 1 | 2
Fluid retention (Metabolism and nutrition disorders) | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0
Nocturia (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.